CLINICAL TRIAL: NCT04508335
Title: Assessment of Effectiveness and Safety of a Novel Pessary for the Non-Surgical Treatment of Pelvic Organ Prolapse
Brief Title: Feasibility Study of the Reia Vaginal Pessary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reia, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-002
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Reia Vaginal Pessary (Experimental)
  Interventions: Device: Reia Vaginal Pessary

INTERVENTIONS:
Device: Reia Vaginal Pessary — Reia Vaginal Pessary

SUMMARY:
The purpose of this study is to obtain preliminary data on the effectiveness, safety, function, comfort, and patient satisfaction with a novel vaginal pessary design for the use in women who suffer from symptoms of pelvic organ prolapse (POP) and have already opted for non-surgical management. Recruited patients will have Stage II POP or greater and will be current users of a Gellhorn or ring style pessary. Following enrollment, each subject will enter a 1-month wash out period in which they will continue using their current pessary so that baseline subjective and objective data can be collected. They will then be fit with a study pessary and enter a 3-month treatment phase. Comparative, subjective, and objective data will be collected at the conclusion of the study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness, safety, function, and comfort of a novel vaginal pessary design for the treatment in women who suffer from of pelvic organ prolapse and who have already opted for non-surgical management. Results will be used to validate prior benchtop testing and to ensure the device performs as anticipated in the real-world environment and does not cause harm. Treatment intervention will be non-blinded to the patient and investigator. Patients will serve as their own controls and enter the treatment phase of the study after a 1-month washout period of using their current pessary. The primary outcome measure will be the change in the scores of the Pelvic Floor Distress Inventory-20 (PFDI-20), administered first during the washout period while still using their current pessary and then at the conclusion of the treatment phase with the study pessary. The PFDI-20 is a validated health-related quality of life instrument to assess the presence and bother of symptoms in women with pelvic floor dysfunction. For women with relatively mild pelvic floor symptoms, a minimal important change (MIC) of between 13.5 and 18.3 points in the PFDI-20 score can be considered clinically relevant. We plan to have at least 40 subjects complete the study. This provides power of .80 for a MIC equivalence limit of 17 points on the PFDI-20 scale. The safety outcome is the prevalence and severity of adverse events that patients experience using the study pessary compared to those experienced with their current pessary. Comparative measurements (in cm) of the most dependent compartment of prolapse in relation to the hymen when using the current and study pessary will be taken to objectively assess function. Comfort will be assessed using a Visual Analogue Scale (VAS - a 10cm linear continuum in which 0 represents no pain and 10 represents worst pain) administered with pessary insertion and removal. Other secondary outcome measures will include global patient satisfaction of the current and study pessary using VAS, percent of patients successfully fit with the study pessary, change in the Pelvic Floor Impact Questionnaire scores between current and study pessary use (the PFIQ is a separate health-related quality of life instrument designed to assess the life impact of pelvic floor symptoms in women with pelvic floor disorders), change in frequency of pessary removal for those patients who insert and remove their pessary outside of medical care (self-managers), and study dropout rates.

The study will take place over 3-4 visits (Visit 0, Visit 1, Visit 2, and Visit 3).

Visit 0 will involve screening, enrollment, and consent. A baseline physical exam will be conducted to assess for pre-existing vaginal adverse events (ecchymoses, abrasions, superficial cuts, erosions, or bleeding) associated with their current pessary use, as well as to assess the ability of their current pessary to support their prolapse by measuring the distance of the most dependent compartment of their prolapse to the hymen. This visit is routinely scheduled for all pessary users and not additional for those consenting to study participation. There will be a washout period where they continue use of their current pessary during which they will complete the PFDI-20, the Pelvic Floor Impact Questionnaire (PFIQ), and the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-IR). Patients who insert and remove their current pessary outside of medical care (self-managers) will track the frequency of removals.

Visit 1 will occur after one month, the conclusion of the washout period. Demographic and historical data will be extracted from the Electronic Medical Record (EMR) and supplemented by the patient as needed. Global patient satisfaction of the current pessary will be assessed using a Visual Analog Scale (VAS). The current pessary will be removed, physical exam will be repeated as in Visit 0, and the presence of perineal disruption associated current pessary removal will be noted. The patient will be fit with the study pessary (which will be used until the study is complete). A VAS will be used to assess the perceived discomfort with removal of the current pessary, and with insertion of the study pessary. For self-managers, teaching will be provided on the proper technique to insert and remove the study pessary and ease of their current pessary removal and reinsertion will be noted using VAS. This visit is additional for those electing to be in the study. A gift card will be offered to compensate for time and travel.

Visit 2 will be scheduled within 1-3 weeks of Visit 1. Visit 2 may be optional at the discretion of the study team. A member of the study team will call the subject ahead of the scheduled Visit 2 to review the subject's experience with the study pessary and adverse events. If the subject has not experienced any complications and the pessary has not dislodged, the study team and subject can decide to omit the in-person Visit 2. The purpose of this visit is to minimize unforeseeable risks associated with use of the study pessary and/or to refit a subject with a study pessary if the original one was expelled or could not be inserted during Visit 1. If Visit 2 occurs in-person, physical exam will be performed to assess for vaginal pathology (ecchymoses, abrasions, superficial cuts, erosions, granulation tissue or bleeding) or urinary retention related to the study pessary, and all adverse events will be recorded. The study pessary will be observed in situ for the presence of rotation and its ability to support prolapse by measuring the distance of the most dependent compartment of the subject's prolapse to the hymen, as well as the distance from the leading edge of the study pessary to the hymen. Those subjects who were not successfully fit with a study pessary in their first visit would be fit with a larger study pessary.

Visit 3 will occur at the conclusion of the 3-month (from Visit 1) treatment phase - a typical length of time between routine visits for patients who choose long term pessary management of their prolapse. When the subject returns for Visit 3, a physical exam will be repeated, as in previous visits, for comparative data. The study pessary will be observed in situ for the presence of rotation and its ability to support prolapse by measuring the distance of the most dependent compartment of the subject's prolapse to the hymen (Points Ba and Bp), as well as the distance from the leading edge of the study pessary to the hymen. A VAS will be used to assess discomfort with removal of the study pessary, discomfort with reinsertion of their current pessary, and their global satisfaction of the study pessary. The subject will have been instructed to return with her current pessary which was removed in Visit 1. If the subject's current pessary is not brought to the visit, she will be given a new pessary of the size and style of her current pessary. Each subject will complete the PFDI-20, PFIQ-7, and PISQ-IR for a post treatment comparison. For self-managers, other data collected will include frequency of removal and a VAS for ease of study pessary insertion and removal.

Specific adverse events (in addition to those described above as part of the physical exam) which will be tracked include pelvic cramping or mild discomfort, bothersome vaginal discharge, urinary tract infection, urinary retention, substantial discomfort, pessary expulsion (deployed or collapsed), pessary failure to deploy or collapse, or adverse event unrelated to the pessary or study visits. Each event will be classified as mild (transient and easily tolerated by the patient), moderate (causing discomfort or interrupting usual activities), or severe (causing considerable interference with usual activities, may be incapacitating, or may require hospitalization). The patient will be instructed to call the triage nursing staff at any point with questions or to report adverse events. The frequency of additional phone calls and any extra visits related to study participation will be tracked. The patient may withdraw from the study and any point upon request.

ELIGIBILITY:
Inclusion Criteria:

* Females with Stage II pelvic organ prolapse or greater
* Users of a Gellhorn or ring style pessary, inclusive of sizes 1.5"-3", for >3 months' duration
* Capable of giving informed consent

Exclusion Criteria:

* Pregnancy Short vaginal length (total vaginal length < 8 cm), or subjective vaginal narrowing
* Deep vaginal erosion noted with removal of current pessary
* Presence of vesicovaginal fistula
* Presence of rectovaginal fistula
* Vaginal, rectal, or bladder tumor
* Presence of open wound or tear near vagina or anus by exam prior to removal of current pessary
* Untreated vaginal or urinary infection requiring treatment
* History of recurrent urinary tract or vaginal infections
* Inflammatory bowel disease
* Chronic pain syndromes of pelvic or anorectal origin
* Previous pelvic floor surgery in last 12 months
* Congenital malformation of bladder, rectum, or vagina
* Significant medical condition interfering with study participation (psychologic, neurologic, active drug/alcohol abuse, etc.)
* Planning pregnancy in next 6 months
* Previous treatment failure with a pessary

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris Strohbehn, MD, Principal Investigator — Dartmouth-Hitchcock Clinic
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Boston Urogynecology Associates, Cambridge, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Medical College, Hawthorne, New York
  - Main Line Health, Media, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - UTHealth, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Reia Pessary: Reia Pessary: Group is fitted with a Reia pessary to manage their pelvic organ prolapse
Period: Overall Study
Arm/Group | Reia Pessary
Started | 78
Treated With Reia Pessary | 62
Completed | 48
Not Completed | 30

BASELINE CHARACTERISTICS:
Population: Demographic information recorded on all enrolled subjects, even those who dropped out before receiving treatment.
Groups:
- Reia Pessary: Reia Pessary: Reia Pessary
Arm/Group | Reia Pessary
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 69
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Floor Distress Inventory-20 (PFDI-20)
Description: The Pelvic Floor Distress Inventory - 20 (PFDI-20) is a validated instrument to assess the presence and bother of symptoms that pelvic floor disorders have on health-related quality of life in women. It is a 20-item questionnaire and the short form of the 46 question PFDI. There are three subscales: Urinary Distress Inventory 6 (UDI-6), Colorectal-Anal Distress Inventory 8 (CRADI-8), and the Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6). The overall score range is 0-300. The higher the score, the greater the perceived impact that pelvic floor dysfunction has on a patient's life. The minimal important change in the PFDI-20 to demonstrate a clinical effect in women choosing conservative management of their prolapse (i.e. a pessary) is between 13.5 and 18.3 points.
Time Frame: At enrollment [Week 0] and post treatment [Week 16]
Population: All subjects treated with the Reia pessary were included in the analysis. Those subjects who withdrew after being treated with the Reia pessary (n = 14) were conservatively considered treatment failures and assigned the upper equivalence limit of 18.3 for the mean different (Reia Pessary - Current Pessary).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Reia Pessary: Reia Pessary: Data from subjects while wearing the Reia pessary
- Current Pessary: Current Pessary: Reia Pessary: Data from subjects while wearing their current pessary
Arm/Group | Reia Pessary | Current Pessary
Number analyzed (Participants) | 48 | 62
score on a scale | 49.46 (43.20) | 62.75 (42.30)
Statistical Analysis 1: Comparison: Reia Pessary; H01: μReia-μCurrent > 18.3 and H02: μReia-μCurrent < -18.3. The alternative hypothesis is thus: HA: -18.3 ≤ μReia-μCurrent ≤ 18.3; Test type: Equivalence — We use 2, one-sided t-tests, each with alpha set at 0.05 to test the composite null hypothesis that the mean difference score (μReia-μCurrent) between the Reia pessary and baseline (current pessary) on the PFDI-20, is greater than 18.3 (H01), the upper equivalence limit, or lower than -18.3 (H02), the lower equivalence limit; p = .0021, t-test, 2 sided

2. Primary Outcome: Adverse Events
Description: Adverse events (AEs) reported by subjects and/or practitioners were recorded and categorized to conform to Common Terminology Criteria for Adverse Events (CTCAE) 5.0 definition. AEs were then categorized into the groups as follows:
  New and/or worsening adverse events: AEs that were not present at baseline with the current pessary but developed with use of the Reia pessary, or that increased in severity with use of the Reia pessary. Improving adverse events: AEs that were present with the current pessary and decreased in severity or were no longer present with use of the Reia pessary. Persisting adverse events: AEs that were present both with the current pessary and with the Reia pessary but did not change in severity.
Time Frame: Throughout study, an average of 16 weeks - AEs may be reported at any time
Measure: Number; unit: participants
Groups:
- Reia Pessary: Reia Pessary: No. of subjects with AE new and/or worsening with Reia pessary
- Current Pessary: Current Pessary: No. subjects experience AE while being treated with their current pessary but improving with Reia pessary
- Persisting Across Pessary Type: No. of subjects with AE persisting across current and Reia pessary
Arm/Group | Reia Pessary | Current Pessary | Persisting Across Pessary Type
Number analyzed (Participants) | 62 | 62 | 62
participants
  Urinary Incontinence | 4 | 2 | 1
  Constipation | 3 | 10 | 3
  Discomfort with Use | 13 | 13 | 10
  Feeling of Obstructed Urination | 2 | 12 | 3
  Granulation Tissue | 14 | 4 | 2
  Sensation of Displacement | 15 | 10 | 10
  Vaginal Abrasions | 12 | 4 | 4
  Vaginal Bleeding | 17 | 4 | 8
  Vaginal Discharge | 18 | 8 | 19
  Vaginal Irritation | 9 | 5 | 2

3. Secondary Outcome: Pelvic Floor Impact Questionnaire (PFIQ-7)
Description: Pelvic Floor Impact Questionnaire-7 is a health-related quality of life instrument, designed to assess the life impact of pelvic floor symptoms in women with pelvic floor disorders. The PFIQ-7 has a parallel structure to the PFDI with 3 Scales: CRAIQ (Colorectal-Anal Impact Questionnaire), POPIQ (Pelvic Organ Prolapse Impact Questionnaire), and IIQ (Incontinence Impact Questionnaire). The PFIQ-7 summary score is calculated by adding the scores of the 3 scales (each range 0 - 100) together (total range 0 - 300). A lower score indicates a lesser life impact of pelvic floor symptoms.
Time Frame: At enrollment [Week 0] and post treatment [Week 16]
Population: Subjects who completed treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reia Pessary
Number analyzed (Participants) | 48
score on a scale
  PFIQ-7 score (current pessary) | 32.23 (49.08)
  PFIQ score (Reia pessary) | 16.86 (21.73)
Statistical Analysis 1: Comparison: Reia Pessary; PFIQ scores at baseline with subjects using current pessary then after treatment with Reia pessary; Test type: Other — Mean difference of PFIQ scores. A negative difference (Reia pessary - current pessary) indicates that the PFIQ-7 score improved with the Reia pessary; p = 0.0192, Wilcoxon (Mann-Whitney) — p value adjusted for multiple variables; Mean Difference (Final Values) = -11.90

4. Secondary Outcome: Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA (International Urogynecological Association)-Revised (PISQ-IR)
Description: A validated evaluation tool which can be used clinically as well as in research for assessment of female sexual function (FSF) in women with female pelvic floor disorders. The PISQ-IR contains 10 sub-scales. The first 4 sub-scales include questions for not sexually active (NSA) people and the following 6 sub-scales include questions for sexually active (SA) people. For not sexually active (NSA) people, higher scores indicate a greater impact of the condition on sexual activity. For sexually active (SA) people, higher scores indicate better sexual function. Transformed sums are reported (0 - 100) for each subscale.
Time Frame: At enrollment [Week 0] and post treatment [Week 16]
Population: Subjects included in this analysis were those that completed the study and had a score for at least 1 sub-scale for both their current pessary and the Reia pessary. Subjects were not required to answer questions regarding their sexual activity to remain in the study. As sexual activity could change during course of the study data for the Reia pessary and current pessary are presented separately, not as a difference.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Current Pessary: Current Pessary: Data from subjects while wearing their current pessary
Arm/Group | Reia Pessary | Current Pessary
Number analyzed (Participants) | 46 | 46
score on a scale
  Not Sexually Active - Partner Related: number analyzed (Participants) | 31 | 31
  Not Sexually Active - Partner Related | 64.0 (32.6) | 58.6 (28.7)
  Not Sexually Active - Condition Specific: number analyzed (Participants) | 31 | 32
  Not Sexually Active - Condition Specific | 24.0 (27.6) | 21.6 (25.9)
  Not Sexually Active - Global Quality: number analyzed (Participants) | 32 | 30
  Not Sexually Active - Global Quality | 28.4 (22.9) | 29.8 (23.8)
  Not Sexually Active - Condition Impact: number analyzed (Participants) | 32 | 30
  Not Sexually Active - Condition Impact | 15.6 (21.5) | 13.7 (22.5)
  Sexually Active - Arousal Orgasm: number analyzed (Participants) | 13 | 14
  Sexually Active - Arousal Orgasm | 68.6 (14.4) | 63.1 (16.7)
  Sexually Active - Condition Specific: number analyzed (Participants) | 13 | 14
  Sexually Active - Condition Specific | 84.5 (24.1) | 94.1 (9.2)
  Sexually Active - Partner Related: number analyzed (Participants) | 12 | 12
  Sexually Active - Partner Related | 76.1 (18.0) | 76.9 (23.4)
  Sexually Active - Desire: number analyzed (Participants) | 13 | 14
  Sexually Active - Desire | 45.4 (14.1) | 44.0 (13.9)
  Sexually Active - Condition Imapct: number analyzed (Participants) | 13 | 14
  Sexually Active - Condition Imapct | 78.8 (26.6) | 76.1 (25.1)
  Sexually Active - Global Quality: number analyzed (Participants) | 13 | 14
  Sexually Active - Global Quality | 69.2 (21.8) | 65.8 (25.4)

5. Secondary Outcome: Objective Assessment of the Pessary's Ability to Support the Prolapse
Description: POP-Q points Ba and Bp will be measured during physical exam, with the pessary in situ. Measurements were averaged to provide one Ba score and one Bp score for each subject for their current pessary and the Reia pessary.
  A more negative number indicates more support of the prolapse (better outcome). Ba ranges from -3 (more support of the prolapse) to 9 (less support of the prolapse). Bp ranges from -3 (more support of the prolapse) to 7 (less support of the prolapse).
Time Frame: At enrollment [Week 0], during treatment [Week 3-5], during treatment [Week 5-7], and at the end of study [Week 16]
Population: A subject's Ba and Bp measurements were included in analysis if the subject had at least 1 data point for both the Reia pessary and their current pessary and did not drop out because of failure to fit.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Current Pessary: Current Pessary: Current Pessary
Arm/Group | Reia Pessary | Current Pessary
Number analyzed (Participants) | 50 | 50
cm
  Ba | -2.14 (0.95) | -1.60 (1.31)
  Bp | -2.32 (0.95) | -2.29 (0.93)

6. Secondary Outcome: Global Assessment of Study Pessary Satisfaction Compared to Current Pessary
Description: Satisfaction will be assessed using a Visual Analog Scale (VAS) with a 100 mm linear continuum in which 0 represents no satisfaction and 100 represents complete satisfaction.
Time Frame: For current pessary at the end of washout period [Week 3-5]; For study pessary post treatment [Week 16]
Population: Only subjects who provided scores for both the current and Reia pessary (including 48 completers and 2 subjects who were treated but did not complete) were included in the analysis group. A negative difference (current pessary - Reia pessary) indicates more satisfaction, i.e., the Reia pessary provides more satisfaction than the current pessary.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Reia Pessary
Number analyzed (Participants) | 50
mm
  Current pessary | 69.68 (24.82)
  Reia pessary | 72.63 (28.02)

7. Secondary Outcome: Pain Associated With Study Pessary Insertion Compared to Current Pessary
Description: Pain will be assessed using a Visual Analog Scale (VAS) with a 100 mm linear continuum in which 0 represents no pain and 100 represents worst pain. Pain scores were averaged to create one pain with insertion of the current pessary and one pain with insertion of the Reia pessary score for each subject.
Time Frame: During treatment [Week 3-5], during treatment [Week 5-7], and post treatment [Week 16]
Population: Subjects' VAS pain scores were included in the analysis group if the subject has at least 1 data point for both the Reia pessary and their current pessary. For each subject with more than one data point, average pain scores for the current pessary and Reia pessary were calculated.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Reia Pessary
Number analyzed (Participants) | 62
mm
  Pain with insertion current pessary | 23.71 (26.58)
  Pain with insertion Reia Pessary | 13.80 (15.82)

8. Secondary Outcome: Pain Associated With Study Pessary Removal Compared to Current Pessary
Description: Pain will be assessed using a Visual Analog Scale (VAS) with a 100 mm linear continuum in which 0 represents no pain and 100 represents worst pain. Pain scores were averaged to create one pain with removal of the current pessary and one pain with insertion of the Reia pessary score for each subject.
Time Frame: During treatment [Week 3-5], during treatment [Week 5-7], and post treatment [Week 16]
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Reia Pessary
Number analyzed (Participants) | 53
mm
  Pain with removal current pessary | 34.27 (30.04)
  Pain with removal study pessary | 23.04 (25.32)

9. Other Pre Specified Outcome: Proportion of Patients Successfully Fit With the Study Pessary
Description: Proportion of patients who were successfully fit with the study pessary.
Time Frame: Post treatment [Week 16]
Population: All subjects who completed the trial were considered successfully fit. For those who did not complete the trial, if the study team indicated that the reason for withdrawal is failure to fit or failure to retain, the subject was considered failed to fit.
Measure: Count of Participants; unit: Participants
Arm/Group | Reia Pessary
Number analyzed (Participants) | 62
Participants
  Subjects success fit | 59
  Fit Failures | 3

10. Other Pre Specified Outcome: Frequency of Pessary Removal for Self-managers
Description: The monthly frequency of pessary self-removal during the washout period will be compared against monthly frequency of self-removal in the treatment phase.
Time Frame: End of washout period (current pessary use before treatment) [Weeks 3-5] and post treatment [Week 16]
Measure: Mean (Standard Deviation); unit: number of times/month
Arm/Group | Reia Pessary
Number analyzed (Participants) | 46
number of times/month
  Self management frequency current pessary | 3.07 (7.36)
  Self management frequency Reia pessary | 2.57 (4.86)

11. Other Pre Specified Outcome: Ease of Insertion of Study Pessary by Subject for Self-managers
Description: Difficulty of insertion was assessed using a visual analog scale (VAS) with a 100 mm linear continuum in which 0 represents very easy and 100 represents very difficult.
Time Frame: End of washout period (current pessary use before treatment) [Weeks 3-5] and post treatment [Week 16]
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Reia Pessary
Number analyzed (Participants) | 33
mm
  Difficulty of insertion current pessary | 33.89 (27.04)
  Difficulty of insertion Reia pessary | 32.79 (25.85)

12. Other Pre Specified Outcome: Ease of Removal of Study Pessary by Subject for Self-managers
Description: Difficulty of removal was assessed using a visual analog scale (VAS) with a 100 mm linear continuum in which 0 represents very easy and 100 represents very difficult.
Time Frame: End of washout period (current pessary use before treatment) [Weeks 3-5] and post treatment [Week 16]
Population: Discrepancy is due to more subjects self-managing the study pessary versus their current pessary.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Reia Pessary
Number analyzed (Participants) | 35
mm
  Difficulty of removal current pessary: number analyzed (Participants) | 33
  Difficulty of removal current pessary | 33.19 (29.14)
  Difficulty of removal Reia pessary | 23.36 (26.42)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 16 weeks
Description: Definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definition. (Non-treatment related Other (Not Including Serious) Adverse Events were not reported in the trial.)
Arm/Group | Reia Pessary | Current Pessary | Persisting Across Pessary Type
All-Cause Mortality (participants affected / at risk) | 1/62 | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/62 | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 51/62 | 55/62 | 55/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reia Pessary (N=62) | Current Pessary (N=62) | Persisting Across Pessary Type (N=62)
Symptomatic coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reia Pessary (N=62) | Current Pessary (N=62) | Persisting Across Pessary Type (N=62)
Vaginal Discharge (Reproductive system and breast disorders) | 18 | 8 | 19
Vaginal Bleeding (Reproductive system and breast disorders) | 17 | 4 | 8 — Vaginal Bleeding
Sensation of Displacement (Reproductive system and breast disorders) | 15 | 10 | 10 — Sensation of displacement of the pessary
Granulation Tissue (Reproductive system and breast disorders) | 14 | 4 | 2 — Vaginal granulation tissue observed during examination
Discomfort with Use (Reproductive system and breast disorders) | 13 | 13 | 10 — Discomfort secondary to use of the pessary
Vaginal Abrasions (Reproductive system and breast disorders) | 12 | 4 | 7
Vaginal Irritation (Reproductive system and breast disorders) | 9 | 5 | 2
Urinary Incontinence (Renal and urinary disorders) | 4 | 2 | 1
Feeling of Obstructed Urination (Reproductive system and breast disorders) | 2 | 12 | 3
Constipation (Reproductive system and breast disorders) | 3 | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT04508335/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT04508335/SAP_001.pdf
  • Informed Consent Form (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT04508335/ICF_002.pdf